CLINICAL TRIAL: NCT04676152
Title: Validation of Noninvasive Blood Pressure Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TORR0004
Record Dates: First submitted 2020-11-05; First posted 2020-12-19 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Hypertension; Hypotension
MeSH Terms: conditions — Hypertension; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test subjects (Experimental): All subjects enrolled had blood pressure measurements taken using the noninvasive blood pressure device.
  Interventions: Device: Masimo Noninvasive Blood Pressure Device

INTERVENTIONS:
Device: Masimo Noninvasive Blood Pressure Device — Non-invasive blood pressure device

SUMMARY:
This is a prospective, nonrandomized multi-center study for the investigation of noninvasive sphygmomanometers.

The purpose of the study is to validate the clinical performance of the Masimo noninvasive blood pressure device compared to reference auscultatory measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Site 1; Stage 1 only: Subjects with a history of hypertension (> 140/85 mmHg) or hypotension (< 100/60 mmHg) within the last 3 months. Stage 2 only: No criterion for blood pressure
* Site 2; Stage 1 and 2: Subjects with systolic blood pressure < 140/90 mmHg.
* Ability to provide informed consent

Exclusion Criteria:

* Febrile subjects
* Subjects displaying respiratory symptoms, or with suspected respiratory illness
* Subjects whose skin is not intact, e.g. wounded, in or at the vicinity of the cuff placement site
* Subjects with removed axillary lymph nodes or mastectomies
* Subjects with peripheral artery disease
* Pregnant women (patient reported)
* Subjects deemed not suitable for the study at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Site 2, Irvine, California
  - Site 1, Lomita, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Subjects: Masimo Noninvasive Blood Pressure Device: All enrolled subjects will have blood pressure measurements done using the Masimo NIBP device and the noninvasive blood pressure device
Period: Overall Study
Arm/Group | Test Subjects
Started | 106
Completed | 97
Not Completed | 9
Not completed — screen fail | 9

BASELINE CHARACTERISTICS:
Arm/Group | Test Subjects
Number analyzed (Participants) | 106
Age, Customized [Count of Participants; unit: Participants]
  Age: <=18 years | 0
  Age: Between 18 and 65 | 88
  Age: >65 years | 15
  Age: Unknown/Not reported | 3
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 59
  Gender: Male | 44
  Gender: Unknown/Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity (NIH/OMB): American Indian or Alaska Native | 0
  Race/Ethnicity (NIH/OMB): Asian | 26
  Race/Ethnicity (NIH/OMB): Native Hawaiian or Other Pacific Islander | 0
  Race/Ethnicity (NIH/OMB): Black or African American | 2
  Race/Ethnicity (NIH/OMB): White | 48
  Race/Ethnicity (NIH/OMB): Hispanic or Latino | 26
  Race/Ethnicity (NIH/OMB): More than one race | 0
  Race/Ethnicity (NIH/OMB): Other | 1
  Race/Ethnicity (NIH/OMB): Unkown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 106

OUTCOME MEASURES:

1. Primary Outcome: Mean and Standard Deviation of Differences Between Masimo NIBP Device and Manual Sphygmomanometer Measurements.
Description: Performance will be determined by calculating the mean and standard deviation of the differences between the systolic and diastolic blood pressure measurements obtained from Masimo NIBP device and manual sphygmomanometer.
Time Frame: 1 hour
Population: Subjects excluded from analysis were as follows:
  * 9 Subjects were screen fails
  * 8 Subjects excluded during data analysis
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Test Subjects
Number analyzed (Participants) | 89
mmHg
  Systolic Blood Pressure | -1.23 (7.32)
  Diastolic Blood Pressure | -2.67 (7.13)

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Test Subjects
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106
Other Adverse Events (participants affected / at risk) | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT04676152/Prot_SAP_000.pdf